CLINICAL TRIAL: NCT04096300
Title: Traditional and Complementary Medicine: a Cure for Idiopathic Granulomatous Mastitis?
Brief Title: An Integrative Approach for Idiopathic Granulomatous Mastitis.
Acronym: IIGM
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Mujgan Calişkan, Professor, Medipol University
Other Study IDs: IMUEC396
Record Dates: First submitted 2019-09-16; First posted 2019-09-19 (Actual); Last update posted 2019-09-19 (Actual); Status verified 2019-09

CONDITIONS: Idiopathic Granulomatous Mastitis
Keywords: Integrative Medicine; Ethnomedicine; Hirudotherapy; Idiopathic Granulomatous Mastitis; Medical Cupping Therapy; Traditional and Complementary Medicine

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples Without DNA — Biopsy Samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Collaboration is established between Turkish Holistic & Integrative Medicine Association and Traditional & Complementary Medicine Society of Istanbul Medipol University.

Study is carried out on idiopathic granulomatous mastitis patients who are followed in the Breast Clinic at Istanbul Medipol University Hospital for between September 2015 and September 2019. Hirudotherapy and medical cupping therapy were applied as traditional and complementary medicine integratively.

Following initial radiological imaging, microbiological- and histological testing, side effects and relapses are analyzed. Follow-up examination is also carried out at the end of the treatment, which consisted of clinical breast exam and radiological imaging.

ELIGIBILITY:
Inclusion Criteria:

* IGM patients, either ones newly diagnosed or had previously received different types of treatments, currently refusing conventional treatments with immunosuppressives etc, or/and surgical management, and now und

Exclusion Criteria:

* Patients currently using any conventional treatment, and/or contraindication to hirudotherapy and cupping.

Ages: 25 Years to 45 Years | Sex: Female
Age Groups: Adult
Study Population: Patients receiving Traditional and Complementary Medicine (T&CM) for IGM will be retrospectively analyzed.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2019-09 (Estimated); Study Completion 2019-09 (Estimated)

PRIMARY OUTCOMES:
Change of Breast Mass Size | Up to 12 months
  Ultrasonic scan at 6 months
Change of Breast Mass Size | Up to 48 months
  Ultrasonic scan at 12 months

SECONDARY OUTCOMES:
Change of Breast Mass Size | Up to 48 months
  MRI scan at 12 months, if prompted by ultrasonic scan

CONTACTS AND LOCATIONS:
Locations (1):
- Medipol University, Beykoz, Istanbul, Turkey (Türkiye)